CLINICAL TRIAL: NCT00363831
Title: A Multi-center Phase II Trial of Capecitabine in Combination With Oxaliplatin (Xelox) as First Line Chemotherapy in Patients With Metastatic Nasopharyngeal Carcinoma (NPC)
Brief Title: Combination of Capecitabine and Oxaliplatin in Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9863
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Oxaliplatin

ARMS (1):
- 1 (Experimental): Oxaliplatin
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — 130mg/m² infusion day 1, repeat every 21 days

SUMMARY:
Primary:

* To evaluate the efficacy of capecitabine in combination with oxaliplatin (XELOX) in terms of overall response rate (based on RECIST criteria) in patients with metastatic NPC without prior chemotherapy for relapse.

Secondary:

* To evaluate the efficacy profile of oxaliplatin (XELOX) in patients with metastatic NPC in terms of time to progression of disease, survival time, duration of response and complete response rate.
* To study the safety and tolerability of the regimen in patients with metastatic NPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed poorly differentiated or undifferentiated nasopharyngeal carcinoma (WHO type II and III) with distant metastasis (ie. other than loco-regional disease). Patients with stage IVc disease, ie. distant metastases on presentation are also eligible.
* Have at least one measurable lesion according to RECIST which has not been irradiated.
* WBC count ≥ 3 x 10^9 /L with neutrophils ≥ 1.5 x 10^9 /L, platelet count ≥ 100 x 10^9 /L and Hb ≥ 9g/dL.
* Serum creatinine ≤ 1.25 ULN
* Be ambulatory and have a Karnofsky Performance Status of ≥ 70% at study entry.
* Recover from prior radiotherapy prior to study entry
* Effective contraception for both male and female if the risk of conception exists.
* Able to swallow and retain oral medication.

Exclusion Criteria:

* Previous cytotoxic chemotherapy for recurrent or metastatic NPC.
* Previous exposure to oxaliplatin and/or capecitabine.
* Pregnant or lactating women. Women of childbearing potential with either positive or no pregnancy test at baseline. Women of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential)
* Sexually active males unwilling to practice contraception during the study.
* Clinically significant cardiac disease (eg. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Patients with a history of central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* Abnormal blood counts, AST, ALT, bilirubin and/or serum creatinine beyond the limits specified in the inclusion criteria.
* Radiotherapy within 4 weeks of treatment start or prior radiotherapy to the indicator lesion(s) being measured in the study (newly arising marker lesions in previously irradiated areas are acceptable).
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Participation in any investigational drug study within 4 weeks preceding the start of treatment.
* Symptomatic peripheral neuropathy NCI-CTCAE grade ≥ 2.
* Known allergic/hypersensitivity reaction to any of the components of study treatments.
* Serious uncontrolled intercurrent infections.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (based on RECIST criteria) | From the beginning to the end of the study

SECONDARY OUTCOMES:
Time to progression | From the beginning to the end of the study
Overall survival time | From the beginning to the end of the study
Adverse events | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Iris Chan, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, Hong Kong, Hong Kong